CLINICAL TRIAL: NCT01034657
Title: A One Year, Open Label, Multicenter Trial of LBH589 Alone or in Combination With ESA in Red Blood Cell Transfusion-dependent LOW and INT-1 MDS Patients Being Either Refractory to ESA or With a Low Probability of Response - the GErman PAnobinostat Low Risk MDS Trial - GEPARD Study
Brief Title: LBH589 Alone or in Combination With Erythropoietin Stimulating Agents (ESA) in Patients With Low or Int-1 Risk Myelodysplastic Syndromes (MDS)
Acronym: GEPARD
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was terminated due to lack of efficacy of single agent LBH589 in the 4 month open label core phase and due to enrollment difficulties.
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLBH589BDE04; EudraCT 2009-010403-84 (Registry Identifier: EudraCT); 2009-010403-84
Record Dates: First submitted 2009-12-16; First posted 2009-12-17 (Estimated); Results first posted 2017-01-25 (Estimated); Last update posted 2017-08-11 (Actual); Status verified 2017-08

CONDITIONS: Myelodysplastic Syndrome (MDS)
Keywords: MDS; bone marrow; anemia; cytopenia; transfusion dependance; EPO; ESA; erythropoietin; LBH589; Myelodysplastic Syndromes; hematopoietic improvement; IPSS Low; IPSS Int-1; HI-E; HDAC Inhibitor; HDAC-I; DAC-I; Deacetylase-Inhibitor; Histone Deacetylase-Inhibitor; red blood cell transfusions
MeSH Terms: conditions — Myelodysplastic Syndromes; Anemia; Cytopenia | interventions — Panobinostat; Epoetin Alfa

ARMS (2):
- LBH589 (Experimental): During the core phase, all participants received oral LBH589 40 mg (30 mg after a protocol amendment) for 4 months. During the randomization phase, participants with hematological improvement of the erythropoetic system (HI-E) and participants with stable disease, who were randomized to single agent LBH589, continued on single agent LBH589 40mg/30mg for an additional 4 months.
  Interventions: Drug: LBH589
- LBH589 + Epoetin Alfa (Experimental): During the randomized phase, participants randomized to LBH589 + Epoetin Alfa (ESA) received oral LBH589 40mg/30mg + ESA 30000 international units (IU)/week injected subcutaneously for 4 months.
  Interventions: Drug: LBH589; Drug: Epoetin Alfa

INTERVENTIONS:
Drug: LBH589 — LBH589 was supplied at dose strengths of 5 mg or 20 mg hard gelatin capsules.
  Other Names: Panobinostat
Drug: Epoetin Alfa — Epoetin alfa was supplied as 10000 IU/1 mL in a ready-to-use syringe.
  Other Names: ESA, HEXAL®
  Arms: LBH589 + Epoetin Alfa

SUMMARY:
This study assessed the efficacy and safety of LBH589 as single agent and in combination with ESA in red blood cell transfusion-dependent Low and Int-1 MDS patients being either refractory to ESA or with a low probability of response. The study had a non-randomized core phase followed by a randomized phase.

ELIGIBILITY:
Key Inclusion Criteria:

* Patients with a lower risk MDS (LOW or INT-1 according to IPSS)
* Red blood cell transfusion dependency of at least 4 Units/8 weeks.
* Not responding to Erythropoietin stimulating agents (ESA) or having a low chance to do so
* Age-adjusted normal cardiac, kidney, liver function

Key Exclusion Criteria:

* Concomitant use of ESA
* Concomitant use of any other investigational drug
* Other malignancy that is not in remission for at least 1 year
* Platelet Count < 75 x 109/L
* Impaired cardiac function or clinically significant cardiac diseases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2009-11; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (12):
- Germany (12):
  - Novartis Investigative Site, Mannheim, Baden-Wurttemberg
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Bonn
  - Novartis Investigative Site, Dresden
  - Novartis Investigative Site, Duisburg
  - Novartis Investigative Site, Düsseldorf
  - Novartis Investigative Site, Frankfurt
  - Novartis Investigative Site, Göttingen
  - Novartis Investigative Site, Hanover
  - Novartis Investigative Site, Leipzig
  - Novartis Investigative Site, München
  - Novartis Investigative Site, Ulm

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was divided into a core phase and a randomized phase. The core phase had an open-label single arm study design. The randomized phase was open-label with two parallel treatment arms for participants with stable disease. Participants with Hematological response of the erythropoietin system remained on single agent oral LBH589.
Pre-assignment Details: Participants with stable disease were eligible for randomization to single agent LBH589 or LBH589 + epoetin alfa. Participants with progressive disease were discontinued. Seven participants who completed the core phase withdrew before the randomization phase.
Groups:
- Not Randomized: Participant, who was eligible for randomization, was not randomized. The participant had stable disease and should have been randomized, but in error, was considered a responder and therefore continued on single agent LBH589.
Period: Core Phase
Arm/Group | LBH589 | LBH589 + Epoetin Alfa | Not Randomized
Started | 34 | 0 | 0
Completed | 20 | 0 | 0
Not Completed | 14 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0
Not completed — Lack of Efficacy | 2 | 0 | 0
Not completed — Abnormal laboratory value | 1 | 0 | 0
Not completed — Adverse Event | 8 | 0 | 0
Not completed — Protocol Violation | 2 | 0 | 0
Period: Randomized Phase
Arm/Group | LBH589 | LBH589 + Epoetin Alfa | Not Randomized
Started | 6 | 6 | 1
Completed | 1 | 0 | 0
Not Completed | 5 | 6 | 1
Not completed — Withdrawal by Subject | 0 | 2 | 0
Not completed — Lack of Efficacy | 5 | 1 | 0
Not completed — Abnormal laboratory value | 0 | 1 | 0
Not completed — Adverse Event | 0 | 2 | 1

BASELINE CHARACTERISTICS:
Population: Core Phase (all participants)
Arm/Group | LBH589
Number analyzed (Participants) | 34
Age, Continuous [Mean (Standard Deviation); unit: Years] | 65.4 (7.70)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 24

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Hematological Response of the Erythropoetic System (HI-E) - Core Phase
Description: HI-E was assessed according to the modified international working group (IWG) criteria for HI. Erythroid response (pretreatment, <11 g/dL): Hgb increase by ≥ 1.5 g/dL, relevant reduction of units of RBC transfusions by an absolute number of at least 4 RBC transfusions/8 wk compared with the pretreatment transfusion number in the previous 8 wk, and only RBC transfusions given for a Hgb of ≤ 9.0 g/dL pretreatment were counted in the RBC transfusion response evaluation; Platelet response (pretreatment, < 100 x 109/L): absolute increase of ≥ 30 x 109/L for participants starting with > 20 x 109/L and platelets Increase from < 20 x 109/L to > 20 x 109/L and by at least 100%; Neutrophil response (pretreatment, < 1.0 x 109/L): at least 100% increase and an absolute increase > 0.5 x 109/L; Progression or relapse after HI: At least 1 of the following: At least 50% decrement from maximum response levels in granulocytes or platelets, reduction in Hgb by ≥1.5 g/dL, or transfusion dependence.
Time Frame: 16 weeks
Population: Participants from the core phase, who had valid response data, were analyzed.
Measure: Number; unit: Percentage of participants
Arm/Group | LBH589
Number analyzed (Participants) | 20
Percentage of participants | 0.0

2. Secondary Outcome: Percentage of Participants With HI-E - Randomized Phase
Description: as for outcome 1
Time Frame: 32 weeks, 52 weeks
Population: Participants from the randomized phase, who had valid response data, were analyzed.
Measure: Number; unit: Percentage of participants
Arm/Group | LBH589 | LBH589 + Epoetin Alfa | Not Randomized
Number analyzed (Participants) | 6 | 6 | 1
Percentage of participants
  32 weeks (n=5,1,1) | 0.0 | 0.0 | 0.0
  52 weeks (n=4,3,1) | 0.0 | 0.0 | 0.0

3. Secondary Outcome: Percentage of Participants With Objective Response During Core Phase
Description: Objective response (complete remission (CR) + partial remission (PR) and HI-platelet (HI-P) response + HI-neutrophil (HI-N) response) was assessed according to the modified IWG criteria: CR bone marrow with 5% myeloblasts with normal maturation of al cell lines (persistent dysplasia is noted) and peripheral blood with Hgb >= 11 g/dL platelets >=100 X 10^9/L, neutrophils >= 1.0 x 10^9/L and blasts 0%. PR = All CR if abnormal before treatment except bone marrow blasts decreased by>=50% over pretreatment but still >5% (ellularity and morphology not relevant). HI-P (pretreatment, < 100 x 109/L) = absolute increase of ≥ 30 x 109/L for participants starting with > 20 x 109/L and platelets Increase from < 20 x 109/L to > 20 x 109/L and by at least 100%; HI-N (pretreatment, < 1.0 x 109/L) = at least 100% increase and an absolute increase > 0.5 x 10^9/L.
Time Frame: 16 weeks
Population: Participants from the core phase, who had valid data, were analyzed.
Measure: Number; unit: Percentage of participants
Arm/Group | LBH589
Number analyzed (Participants) | 20
Percentage of participants | 0.0

4. Secondary Outcome: Percentage of Participants With Objective Response During the Randomized Phase
Description: as for outcome 3
Time Frame: 32 weeks, 48 weeks
Population: Participants from the randomized phase, who had valid data, were analyzed.
Measure: Number; unit: Percentage of participants
Arm/Group | LBH589 | LBH589 + Epoetin Alfa | Not Randomized
Number analyzed (Participants) | 6 | 6 | 1
Percentage of participants
  Week 32 ( n=5,1,1) | 0.0 | 0.0 | 0.0
  Week 48 (n=6,5,1) | 0.0 | 0.0 | 0.0

5. Secondary Outcome: Frequency Distribution of IPSS Score Status - Core Phase
Description: The IPSS score values were calculated based on the results of bone marrow analysis. A score value of 0 has bone marrow blast <5%, karyotype of normal, sole: -Y, del 5Q, del 20q and cytopenias (lineages affected) of 0 to 1. Score value of 0.5 has 5-10 bone marrow blasts, karyotype of Others and cytopenias of 2 to 3. A score value of 1.0 has complex >= 3 chromosomal abnormalities and/or chromosome 7 anomalies. A score of 1.5 has 11-20 bone marrow blasts and a score of 2.0 has 21-30 bone marrow blasts. The prognostic score is determined by the sum of the single scoring values. The risk groups are determined as follows: Low = 0 points (5.7 years of median survival); intermediate -1 (INT-1) = 0.5-1.0 points (3.5 years of median survival); INT-2 = 1.5-2.0 points (1.2 years of median survival); and high >=2.5 points (6 months of median survival).
Time Frame: baseline
Population: All participants from the core phase were analyzed.
Measure: Number; unit: Percentage of participants
Arm/Group | LBH589
Number analyzed (Participants) | 34
Percentage of participants
  Baseline (core phase), Low | 32.4
  Baseline (core phase),, INT-1 | 67.6
  Baseline (core phase),, INT-2 | 0.0
  Baseline (core phase), High | 0.0

6. Secondary Outcome: Frequency Distribution of IPSS Score Status - Randomized Phase
Description: as for outcome 5
Time Frame: 52 weeks
Population: Only participants from the randomized phase, who had values at week 52, were included in the analysis.
Measure: Number; unit: Percentage of participants
Arm/Group | LBH589 | LBH589 + Epoetin Alfa | Not Randomized
Number analyzed (Participants) | 6 | 6 | 1
Percentage of participants
  Week 52 (randomized phase), Low | 0.0 | 0.0 | 100.0
  Week 52 (randomized phase), , INT-1 | 16.7 | 16.7 | 0.0
  Week 52 (randomized phase), INT-2 | 0.0 | 0.0 | 0.0
  Week 52 (randomized phase), HIgh | 0.0 | 0.0 | 0.0

7. Secondary Outcome: Mean Single Scoring Values of the IPSS - Core Phase
Description: as for outcome 5
Time Frame: baseline
Population: All participants from the core phase were analyzed.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | LBH589
Number analyzed (Participants) | 34
units on a scale | 0.43 (0.351)

8. Secondary Outcome: Mean Single Scoring Values of the IPSS - Randomized Phase
Description: as for outcome 5
Time Frame: 52 weeks
Population: Participants from the randomized phase, who had values at week 52, were included in the analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | LBH589 | LBH589 + Epoetin Alfa | Not Randomized
Number analyzed (Participants) | 1 | 1 | 1
units on a scale | 1.0 (NA) — Standard deviation cannot be calculated because only 1 participant was analyzed. | 1.0 (NA) — Standard deviation cannot be calculated because only 1 participant was analyzed. | 0.0 (NA) — Standard deviation cannot be calculated because only 1 participant was analyzed.

9. Secondary Outcome: Overall Survival (OS) - Overall Period
Description: OS was defined as the time from start of treatment to death from any cause.
Time Frame: 48 weeks
Population: All participants from the core phase were analyzed.
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | LBH589
Number analyzed (Participants) | 34
months | NA [NA to NA] — The median could not be calculated because only 1 event occurred.

10. Secondary Outcome: Time to Response - Overall Period
Description: Time to response was defined as the time from start of treatment to the first documented response (complete [CR] or partial [PR]) according to modified IWG criteria for HI.
Time Frame: 52 weeks
Population: Time to response could not be evaluated because there was no response.
Arm/Group | LBH589 | LBH589 + Epoetin Alfa | Not Randomized
Number analyzed (Participants) | 0 | 0 | 0

11. Secondary Outcome: Event-free Survival (EFS) - Overall Period
Description: EFS was defined as the time from start of treatment to failure or death from any cause.
Time Frame: 52 weeks
Population: Event-free survival could not be evaluated because there was no response, no progression or no disease-free period.
Arm/Group | LBH589 | LBH589 + Epoetin Alfa | Not Randomized
Number analyzed (Participants) | 0 | 0 | 0

12. Secondary Outcome: Progression-free Survival (PFS) - Overall Period
Description: PFS was defined as the time from start of treatment to disease progression or death from MDS.
Time Frame: 52 weeks
Population: PFS could not be evaluated because there was no progression.
Arm/Group | LBH589 | LBH589 + Epoetin Alfa | Not Randomized
Number analyzed (Participants) | 0 | 0 | 0

13. Secondary Outcome: Disease-free Survival (DFS) - Overall Period
Description: DFS was defined as the time from start of treatment to the time to relapse.
Time Frame: 52 weeks
Population: DFS could not be evaluated because there was no disease-free period.
Arm/Group | LBH589 | LBH589 + Epoetin Alfa | Not Randomized
Number analyzed (Participants) | 0 | 0 | 0

14. Secondary Outcome: Time to Cause-specific Death - Overall Period
Description: Time to cause-specific death was defined as the time from start of treatment to death related to MDS.
Time Frame: 52 weeks
Population: Time to cause-specific death could not be evaluated because there was no cause-specific death.
Arm/Group | LBH589 | LBH589 + Epoetin Alfa | Not Randomized
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Groups:
- LBH589 - Core Phase: During the core phase, all participants received oral LBH589 40 mg (30 mg after a protocol amendment) for 4 months. During the randomization phase, participants with hematological improvement of the erythropoetic system (HI-E) and participants with stable disease, who were randomized to single agent LBH589, continued on single agent LBH589 40mg/30mg for an additional 4 months.
- LBH589 - Randomized Phase; LBH589 + ESA - Randomized Phase: During the randomized phase, participants randomized to LBH589 + Epoetin Alfa (ESA) received oral LBH589 40mg/30mg + ESA 30000 international units (IU)/week injected subcutaneously for 4 months.
Arm/Group | LBH589 - Core Phase | LBH589 - Randomized Phase | LBH589 + ESA - Randomized Phase | Not Randomized
Serious Adverse Events (participants affected / at risk) | 11/34 | 1/6 | 1/6 | 1/1
Other Adverse Events (participants affected / at risk) | 34/34 | 6/6 | 6/6 | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | LBH589 - Core Phase (N=34) | LBH589 - Randomized Phase (N=6) | LBH589 + ESA - Randomized Phase (N=6) | Not Randomized (N=1)
Coronary artery stenosis (Cardiac disorders) | 1 | 0 | 0 | 0
Myocardial infarction (Cardiac disorders) | 1 | 0 | 0 | 0
Sudden hearing loss (Ear and labyrinth disorders) | 1 | 0 | 0 | 0
Optic ischaemic neuropathy (Eye disorders) | 0 | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Faecaloma (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Chest pain (General disorders) | 1 | 0 | 0 | 0
Impaired healing (General disorders) | 1 | 0 | 0 | 0
Pyrexia (General disorders) | 1 | 0 | 0 | 0
Abscess limb (Infections and infestations) | 0 | 0 | 1 | 0
Lymph node abscess (Infections and infestations) | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 0 | 0
Postoperative wound infection (Infections and infestations) | 1 | 0 | 0 | 0
Sepsis (Infections and infestations) | 1 | 0 | 0 | 0
Septic shock (Infections and infestations) | 1 | 0 | 0 | 0
Staphylococcal infection (Infections and infestations) | 0 | 0 | 1 | 0
Subcutaneous abscess (Infections and infestations) | 0 | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Chronic myelomonocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Glomerulonephritis (Renal and urinary disorders) | 1 | 0 | 0 | 0
Haematuria (Renal and urinary disorders) | 1 | 0 | 0 | 0
Urinary incontinence (Renal and urinary disorders) | 1 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Phlebitis (Vascular disorders) | 0 | 0 | 1 | 0
Vascular pseudoaneurysm (Vascular disorders) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | LBH589 - Core Phase (N=34) | LBH589 - Randomized Phase (N=6) | LBH589 + ESA - Randomized Phase (N=6) | Not Randomized (N=1)
Anaemia (Blood and lymphatic system disorders) | 3 | 1 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 4 | 1 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 12 | 1 | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 14 | 1 | 1 | 0
Vertigo (Ear and labyrinth disorders) | 5 | 0 | 0 | 0
Hypothyroidism (Endocrine disorders) | 6 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 3 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 3 | 1 | 0 | 0
Cheilitis (Gastrointestinal disorders) | 2 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 3 | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 24 | 1 | 3 | 0
Dyspepsia (Gastrointestinal disorders) | 5 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 18 | 1 | 1 | 0
Stomach discomfort (Gastrointestinal disorders) | 2 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 2 | 0 | 0 | 0
Teeth brittle (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 9 | 1 | 0 | 0
Asthenia (General disorders) | 7 | 0 | 0 | 0
Fatigue (General disorders) | 16 | 1 | 0 | 0
Gait disturbance (General disorders) | 0 | 1 | 0 | 0
Influenza like illness (General disorders) | 0 | 1 | 0 | 0
Oedema peripheral (General disorders) | 2 | 3 | 1 | 0
Pyrexia (General disorders) | 2 | 0 | 0 | 0
Hypersensitivity (Immune system disorders) | 2 | 0 | 0 | 0
Abdominal wall abscess (Infections and infestations) | 0 | 0 | 0 | 1
Bronchitis (Infections and infestations) | 2 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 3 | 1 | 1 | 0
Urinary tract infection (Infections and infestations) | 2 | 1 | 0 | 0
Post procedural haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Transfusion reaction (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Blood bilirubin increased (Investigations) | 1 | 1 | 0 | 0
Blood creatinine increased (Investigations) | 2 | 0 | 1 | 0
Blood iron increased (Investigations) | 0 | 1 | 0 | 0
Blood thyroid stimulating hormone increased (Investigations) | 3 | 0 | 0 | 0
Weight decreased (Investigations) | 8 | 3 | 0 | 0
Anorexia (Metabolism and nutrition disorders) | 9 | 0 | 0 | 0
Haemochromatosis (Metabolism and nutrition disorders) | 3 | 0 | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 2 | 0 | 0 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 2 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 2 | 1 | 1
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 5 | 0 | 2 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 4 | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Dysgeusia (Nervous system disorders) | 4 | 0 | 0 | 0
Headache (Nervous system disorders) | 3 | 0 | 0 | 0
Depression (Psychiatric disorders) | 0 | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 4 | 0 | 0 | 0
Skin fissures (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1
Haematoma (Vascular disorders) | 2 | 1 | 0 | 0
Hypertension (Vascular disorders) | 1 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety.